CLINICAL TRIAL: NCT06547060
Title: Leggings With Resistance Bands on Caloric Expenditure During Exercise
Status: Not yet recruiting | Type: Observational
Sponsor: University of Texas at Austin (Other)
Collaborators: Sweetflexx Resistance Activewear (Unknown)
Responsible Party: Sponsor
Other Study IDs: STUDY00005845
Record Dates: First submitted 2024-07-26; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Health Behavior
Keywords: Fat oxidation; Energy expenditure; Post-exercise oxygen consumption; Healthy female; Shortened resistance leggings; Cardiovascular response; Metabolic response; moderate to high intensity; Calorie expenditure
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cross-over self-control group: The current study utilizes the cross-over design. Therefore, only one group of participants will be studied using the self-control design. Each participant will undergo two conditions (control leggings vs. shortened resistance band leggings) at least one day apart.
  Interventions: Other: Exercise leggings

INTERVENTIONS:
Other: Exercise leggings — The participants will wear two types of leggings (i.e., control leggings vs. leggings with shortened resistance bands) while performing the same exercise on two different days, respectively.

SUMMARY:
The primary aim of this study is to investigate the impact of incorporating shortened resistance bands (SRB) into leggings on cardiovascular responses and caloric expenditure during exercise in young, healthy women. This study will employ a randomized, controlled, and double-blind crossover design involving four types of exercise: walking, climbing, rowing, and cycling. Participants will perform each type of exercise for 10 minutes while wearing either SRB leggings or leggings without SRB, with sessions on separate days and about 3 days apart. The cardiovascular and metabolic responses will be measured during and after the exercise.

DETAILED DESCRIPTION:
This study will employ a randomized, controlled, and single-blind crossover design involving stair climbing, rowing, and cycling exercises for 10 minutes while wearing either SRB leggings or leggings without SRB (control leggings) on separate days (with at least three days in between). The goal is to compare the metabolic and cardiovascular responses of exercising with different types of leggings.

Participants will be randomly assigned to wear either SRB leggings or control leggings first and then switch to the other type of leggings for the exercise testing on a separate day. The sequence of exercises will also be randomized for each participant but will remain consistent for each participant. The participants, technicians, and PIs will be blinded as to which type of leggings were used on a given day, with leggings being coded as "A" or "B" and provided prelabeled by SweetflexxTM company.

The study will consist of three laboratory visits:

1. Laboratory visit 1 (Visit 1): Screening, informed consent, health-related questionnaires, familiarization, exercise pace determination, and legging size fitting. This visit will take 1 hour.
2. Laboratory visit 2 (Visit 2): Walk on the treadmill, climb on the StairMaster, row on a rowing ergometer, and cycle on a bicycle ergometer with one type of leggings. This visit will take 2 hours.
3. Laboratory visit 3 (Visit 3): Repetition of walking on the treadmill, climbing on the inclined StairMaster, rowing on a rowing ergometer, and cycling on a bicycle ergometer with another type of leggings. This visit will take 2 hours.

Exercise sessions

Exercise pace determination and familiarization procedures (Visit 1). Each participant will perform the identical exercises on the StairMaster (Matrix, Cottage Grove, WI, USA), rowing ergometer (Concept II, Morrisville, VT, USA), and cycle ergometer (Lode, Groningen, Netherlands) on separate days. Because participants may not have experience with the exercise equipment used in this study, they will be thoroughly trained and familiarized with all exercise maneuvers and routines after screening and informed consent processes to ensure comfort and consistency. The exercise pace for each piece of equipment will be chosen during familiarization based on the participant's ability to maintain each type of exercise for at least 10 minutes. This pre-exercise testing stage will standardize the exercise parameters for each piece of equipment and allow participants to familiarize themselves with them. Parameters of pace standardization will include walking speed (mph) for the treadmill, climbing speed (steps/minute) and incline level for StairMaster, stroke output (watts) and rowing speed (strokes/minute) for the rowing ergometer, and revolutions per minute and workload (watts) for the bicycle ergometer. The exercise pace for each piece of equipment will be standardized between the two testing days. This stage will take 5 minutes for each exercise equipment, with a 5-minute rest between each type of exercise.

Climbing, rowing, and cycling exercise tests (Visit 2 and 3). Participants will have two laboratory visits for exercise testing scheduled at the same time of day. Upon arrival at the laboratory, participants will change into control or SRB leggings according to the randomization. This randomization will be conducted through a mobile application randomizer. They will then be weighed and equipped with a heart rate monitor (Polar®, Kempele, Finland) and a digital blood pressure monitor (Omron Corp., Kyoto, Japan). Participants will rest for 10 minutes in a quiet room in a sitting position, followed by the measurement of heart rate and blood pressure. After 5 minutes of exercise, participants will wear a face mask (Hans Rudolph Inc., Kansas, America) for metabolic testing connected to a calibrated metabolic cart to collect the inhaled and exhaled air during exercise.

Each exercise session will last 10 minutes, with the first 5 minutes acclimating to the exercise and the remaining 5 minutes as steady-state exercise. Therefore, data from the last 5 minutes will be used to analyze energy expenditure. If a participant cannot reach a steady state within the first 5 minutes, the exercise will continue until 5 minutes after reaching the steady state. A steady state is defined as the point at which oxygen consumption (VO2) plateaus during submaximal aerobic exercise (2). It is typically reached within 1-4 minutes under the maintained and submaximal exercise intensity (2, 3). The purpose of achieving a steady state is to measure caloric expenditure.

After each type of exercise, participants will quickly move to the seated position in a standardized chair with the face mask on to continuously measure the post-exercise metabolic response. They will rest for 10 minutes to ensure their heart rate and blood pressure return to normal before the next exercise session. To better standardize the rowing exercise on two exercise testing days, participants will start at full knee flexion and end at full leg extension during each stroke of the rowing exercise. A metronome will be used to standardize the frequency of the rowing stroke.

Measurements

Anthropometric measures. Before the start of the exercise, participants' height, body weight, and body composition will be measured noninvasively through a bioimpedance device (Tanita Corp., Tokyo, Japan) will be measured. Various circumferences will be recorded, including abdominal circumference across the umbilicus, hip circumference at the widest part of the buttocks, thigh circumference at the midpoint between the hip bone and mid-patella, and calf circumference at the widest part. These measurements will be conducted by the same investigator to ensure consistency, and each circumference measurement will be taken at least twice, with the average value used for analysis.

Cardiovascular responses. Heart rate will be monitored continuously throughout the whole test by a heart rate sensor (Polar®, Kempele, Finland). Systolic, diastolic, and mean blood pressures will be measured in the right arm positioned at heart level with a digital blood pressure monitor (Omron Corp., Kyoto, Japan) before and every two minutes after each type of exercise until the blood pressure recovers back to baseline. Rating of perceived exertion (RPE) will be asked every two minutes during the exercise until the completion of every exercise session, with 6 representing resting and 20 indicating maximal effort.

Metabolic responses. Oxygen consumption (VO2) and carbon dioxide production (VCO2), along with the respiratory exchange ratio (RER = VCO2/VO2), will be measured using a calibrated metabolic cart (TrueOne®, Salt Lake City, UT, USA). Respiratory exchange ratio (RER) and VO2 values during a 5-minute steady state will be used to calculate caloric expenditure (kcal) and fat oxidation using the indirect calorimetry method. All metabolic responses will be continuously monitored throughout the whole session.

Core temperature. The core temperature (℃) will be measured before and after each type of exercise using a tympanic thermometer to detect the temperature from the tympanic membrane. This method is a simple and safe way to measure core temperature.

Questionnaires and surveys

Physical Activity Readiness Questionnaire (PAR-Q+) and Laboratory Health Research Questionnaire. The PAR-Q is a simple self-screening tool that is typically used by fitness trainers or coaches to determine the safety or possible risks of exercising based on health history, current symptoms, and risk factors. It will be utilized to determine the participants' eligibility for exercise testing (see appendix). Participants will complete a health questionnaire developed by our laboratory, providing information on self-medical history, family medical history, medication, alcohol and smoking habits, and physical activity. This will be done on paper, cell phones, or a tablet according to their preference after obtaining their informed consent. The electronic version is supported by the Qualtrics system (https://utexas.qualtrics.com/jfe/form/SV_781SzF02Ak1nCsu).

Female research health questionnaire. In Visit 1, participants will also complete a female health research questionnaire adapted from the questionnaire developed by the Bruno Balke Biodynamics Laboratory at the University of Wisconsin (see appendix). This questionnaire covers menstruation history, contraceptive use, contraceptive history, and pregnancy history. The purpose of this questionnaire is to gather information on the menstrual cycle for each participant, which will be used to standardize the menstrual cycle phase on the two exercise testing days for each participant.

Leggings evaluation questionnaire. At the conclusion of the testing session, the participants will complete the legging evaluation survey. This questionnaire evaluates the comfort and compression sensation or limitation in various regions of the leggings, including the waist, hip, crotch area, thigh, and calf. Providing additional positive and negative feedback is optional.

Environmental controls

Experimental setting control. All exercise tests will be conducted at a temperature of 25°C. Before the exercise testing, participants should fast for at least 4 hours (water is allowed), refrain from caffeine consumption for 12 hours before coming in, avoid alcohol and strenuous exercise for 24 hours before testing, and get adequate sleep.

Physical activity and diet control. The participants will maintain their normal diet and level of activity for 24 hours before the experimental protocols in Visit 2. They will complete a 24-hour exercise and dietary recall. According to the previous recall, participants will be asked to repeat their diet and exercise 24 hours before Visit 3. They will be asked to maintain their normal diet and physical activity before completing all lab visits.

Menstrual cycle control and contraceptives control. The menstrual cycle has been shown to have a small but significant effect on energy expenditure, metabolic rate, and body temperature, although recent evidence showed conflicting results. To control for this confounding factor, each participant's testing will be scheduled in the same menstrual cycle phases. (i.e., two exercise test days are either at the middle luteal or early follicular phases). These two phases have relatively stable sex hormone levels throughout the menstrual cycle. Participants who are taking oral contraceptive medication will be recommended to maintain the same medication regimen on exercise testing days. Participants will be encouraged to use barrier contraception during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young to middle-aged women
* Body mass index (BMI) ranging from 18.5 to 35 kg/m²
* Physical activity level of ≤ 3 sessions of moderate to vigorous exercise per week

Exclusion Criteria:

* Pregnancy or lactation
* Alcohol abuse
* Musculoskeletal joint issues that could affect exercise performance
* Contraindications to exercise (e.g., recent myocardial infarction)
* Current COVID-19 diagnosis
* Current smoker
* Overt cardiovascular disease
* Use of medications that might affect the cardiovascular or metabolic system (e.g., hormone replacement therapy)
* Non-English speaker

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be non-smoking, healthy, young to middle-aged women of all races and ethnic backgrounds. The proposed study includes exclusively female participants because the targeted leggings are specifically designed for women.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Calorie expenditure in kilocalories (kcal) | The oxygen consumption will be monitored during four 10-minute exercises (i.e., rowing, walking, climbing and cycling) and the 10-minute recovery period following the completion of each 10-minute exercise.
  Oxygen consumption values will be used to calculate caloric expenditure (kcal) and fat oxidation (kcal) using the indirect calorimetry method.
Fat oxidation in kilocalories (kcal) | The oxygen consumption and respiratory exchange ratio will be monitored during four 10-minute exercises (i.e., rowing, walking, climbing and cycling) and the 10-minute recovery period following the completion of each 10-minute exercise.
  Respiratory exchange ratio (RER) and oxygen consumption values will be used to calculate fat oxidation (kcal) using the indirect calorimetry method.

SECONDARY OUTCOMES:
Heart rate in beats per minute (bpm) | Heart rate will be monitored at baseline, during four 10-minute exercises (i.e., rowing, walking, climbing and cycling), and the 10-minute recovery period following the completion of each 10-minute exercise.
  Heart rate is the number of heart beat per minute (bpm).
Blood pressure in millimeters of mercury (mmHg) | Systolic blood pressure and diastolic blood pressure will be monitored at baseline and every two minutes during the 10-minute recovery period following each 10-minute exercise (i.e., rowing, walking, climbing and cycling, respectively).
  Both systolic blood pressure and diastolic blood pressure will be measured.
Rate of perceived exertion | RPE will be measured every minute during four 10-minute exercises (i.e., rowing, walking, climbing and cycling).
  Rate of perceived exertion (RPE) is a subjective measure to indicate the participant's feeling about the exercise.
Core temperature in Celsius (°C) | The core temperature will be measured at baseline and every two minutes during 10-minute recovery period following each 10-minute exercise (i.e., rowing, walking, climbing and cycling, respectively).
  The core temperature will be measured in the ear by using a digital ear thermometer.
Leggings evaluation | Participants will fill out a leggings evaluation survey immediately after the last 10-minute recovery period following the completion of the fourth/last 10-minute exercise bout.
  The participant will fill out a survey on their feeling about exercising with each type of leggings, including their previous leggings-wearing experience and satisfaction level with tested leggings.

CONTACTS AND LOCATIONS:
Overall Officials: Hirofumi Tanaka, Ph.D., Principal Investigator — The University of Texas at Austin
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Identifiable data will only be available to the research team members involved in the project (i.e., the PI and research assistants) and sponsors upon request. Depending on the scientific journals to which we submit this research, de-identified data may be shared with other investigators upon reasonable request, as data availability has become an important element in scientific publications.